CLINICAL TRIAL: NCT01425268
Title: AirXpanders Patient Activated Controlled Tissue Expander System for Breast Reconstruction
Brief Title: Patient Controlled Tissue Expansion for Breast Reconstruction
Acronym: XPAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AirXpanders, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP-0003 AirXpanders
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: Tissue Expansion; Tissue Expander; Breast Tissue Expansion; Breast Tissue Expander; Breast Reconstruction; Two Stage Breast Reconstruction; 2 Stage Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms | interventions — Tissue Expansion Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (2):
- AeroForm Tissue Expansion (Experimental): AeroForm Tissue Expansion inflation with carbon dioxide by remote control
  Interventions: Device: AeroForm Tissue Expansion
- Saline Tissue Expansion (Active Comparator): Saline Tissue Expansion inflated by needle injections of saline
  Interventions: Procedure: Saline Tissue Expansion

INTERVENTIONS:
Device: AeroForm Tissue Expansion — The AeroForm Patient Controlled Tissue Expander is a breast tissue expander implanted following mastectomy and activated by remote control to release small doses of carbon dioxide from an internal reservoir to fill and inflate the expander.
  Other Names: AirXpander Tissue Expander System; Patient Activated Controlled Expansion (PACE); AeroForm Patient Activated Tissue Expander; AeroForm Tissue Expander System; AeroForm Tissue Expander
  Arms: AeroForm Tissue Expansion
Procedure: Saline Tissue Expansion — A saline tissue expander is a breast tissue expander which is implanted following mastectomy and inflated over time using needle injections to fill and inflate the expander with saline.
  Other Names: saline breast tissue expander; saline expander; breast tissue expander; tissue expander
  Arms: Saline Tissue Expansion

SUMMARY:
This study is designed to compare the performance and safety of the AirXpander tissue expander to standard saline expanders in patients undergoing two-stage breast reconstruction following mastectomy.

DETAILED DESCRIPTION:
This is a pivotal, prospective, multi-center randomized, controlled, open-label clinical study designed to compare the performance and safety of the AirXpander Tissue Expander System to currently cleared saline tissue expanders. Subject who meet the inclusion and agree to participate in the study will be enrolled and randomized to either the investigational arm (AirXpander Tissue Expander) or the control arm (standard saline tissue expander) using a 2:1 (AirXpander to saline) permuted block randomization stratified by investigational center and procedure (unilateral or bilateral). If the subject is having a bilateral procedure, the same type of expander will be implanted in each side. Subjects in both arms will be followed in the same manner until the explantation of the tissue expander(s) and exchange for permanent implant(s).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a woman between the ages of 18-70.
2. Subject needs to have tissue expansion as part of her breast reconstruction.
3. Subject is able to provide written informed consent.
4. Subject is able and willing to comply with all of the study requirements.
5. Subject is able to understand and manage at home dosing regimen.

Exclusion Criteria:

1. Subjects skin is not suitable for tissue expansion.
2. Subject has remaining tumor cells following her mastectomy.
3. Subject has a current or prior infection at the intended expansion site.
4. Subjects skin has been damaged by previous radiation treatments and the use of non radiated tissue from another part of her body will not be used.

4a. Subject had planned radiation therapy at the intended expansion site while the expander is implanted.

5. Subject has a history of failed tissue expansion or breast implantation at the intended expansion site.

6. Subject has any existing medical condition that the doctor thinks puts the subject at an increased risk of complications (e.g., severe collagen vascular disease, poorly managed diabetes).

7. Subject is taking any medications that the doctor thinks puts the subject at an increased risk of complications (e.g., prednisone, Coumadin).

8. Subject is currently participating in a concurrent investigational drug or device study.

9. Subject is a current tobacco smoker. 10. Subject is overweight (BMI > 33). 11. Subject is unwilling to comply with the air travel or altitude restriction of not > 3300 feet (1000 meters) from baseline during the time the AeroForm tissue expander is implanted.

12. Subject has a currently implanted electronic device such as a pacemaker, defibrillator, neurostimulator device, or drug infusion device.

13. Subject is pregnant or planning on becoming pregnant during the study period.

14. Subject has a history of psychological condition, drug or alcohol misuse which may interfere with their ability to use the device safely.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2011-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Ascherman, M.D., Principal Investigator — New York-Presbyterian Hospital / Columbia University
Locations (17):
- United States (17):
  - Marin General Hospital, Greenbrae, California
  - Susan Downey, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Sutter Healthcare-Sacramento, Sacramento, California
  - Good Samaritan Hospital, San Jose, San Jose, California
  - eSSe Plastic Surgery, Fort Lauderdale, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Norton Healthcare Pavilion, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Columbia University, New York, New York
  - South Nassau Communities Hospital, Oceanside, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ascherman JA, Zeidler K, Morrison KA, Appel JZ, Berkowitz RL, Castle J, Colwell A, Chun Y, Johnson D, Mohebali K. Carbon Dioxide-Based versus Saline Tissue Expansion for Breast Reconstruction: Results of the XPAND Prospective, Randomized Clinical Trial. Plast Reconstr Surg. 2016 Dec;138(6):1161-1170. doi: 10.1097/PRS.0000000000002784. PMID 27879582
- [Derived] Zeidler KR, Berkowitz RL, Chun YS, Alizadeh K, Castle J, Colwell AS, Desai AR, Evans G, Hollenbeck S, Johnson DJ, Morris D, Ascherman JA. AeroForm patient controlled tissue expansion and saline tissue expansion for breast reconstruction: a randomized controlled trial. Ann Plast Surg. 2014 May;72 Suppl 1:S51-5. doi: 10.1097/SAP.0000000000000175. PMID 24740025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited were current patients at the investigator's practice who were scheduled to undergo two-stage breast reconstruction between November 2011 - December 2014.
Period: Overall Study
Arm/Group | AeroForm Tissue Expansion | Saline Tissue Expansion
Started | 106 (106 Subjects Randomized to AeroForm Arm / 98 Subjects Treated (Implanted)) | 52 (52 Subjects Randomized to Saline Arm / 52 Subjects Treated (Implanted))
Completed | 98 | 52
Not Completed | 8 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Sponsor Decision | 5 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AeroForm Tissue Expansion | Saline Tissue Expansion | Total
Number analyzed (Participants) | 98 | 52 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 92 | 49 | 141
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (9.83) | 51.1 (9.88) | 49.7 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 52 | 150
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 98 | 52 | 150

OUTCOME MEASURES:

1. Primary Outcome: Successful Tissue Expansion and Exchange to a Permanent Breast Implant Unless Precluded by a Non-device Related Event
Description: The primary endpoint is assessed when the subject has completed tissue expansion and completed an exchange to standard breast implants. Subjects not completing the exchange procedure due to a device related event are considered failures.
Time Frame: 12 months
Population: Primary Analysis Population (Per Protocol Cohort) = Subjects with an expander implanted successfully with no major protocol violation (evaluated per breast). Subjects who had a bilateral procedure have each breast evaluated separately.
Measure: Count of Units; unit: Breasts
Units Other Than Participants: Breasts
Arm/Group | AeroForm Tissue Expansion | Saline Tissue Expansion
Number analyzed (Participants) | 98 | 52
Number analyzed (Breasts) | 155 | 83
Breasts | 149 | 82
Statistical Analysis 1: Comparison: AeroForm Tissue Expansion vs Saline Tissue Expansion; The study was powered to show that the Treatment Success rate for the AeroForm System (πTreatment) was not worse than the rate for the saline expander (πControl) by more than 10% (-0.10 < πTreatment - πControl); Test type: Non-Inferiority — Assuming that the success rate for both expanders was 95%, at least 92 breasts implanted with a AeroForm Tissue Expander and 46 breasts implanted with a saline expander were needed to be 80% confident (i.e., have a statistical power of 80%) that the lower bound of the one-sided 95% Confidence Interval for the difference in the Success rates (πTreatment - πControl) was greater than or equal to -10%; margin of non-inferiority = -7.3, 95% CI 1-sided [lower limit -7.3241] — The Treatment Success Rate per breast is 96.1% (149/155) for AeroForm and 98.8% (82/83) for saline.The difference (AeroForm - saline) is -2.7% with a lower confidence limit of -7.3%, meeting the non-inferiority margin of > -10%

2. Secondary Outcome: Expansion Days
Description: The median number of days taken to complete the expansion process.
Time Frame: 12 months
Population: All breasts successfully exchange from expander to standard breast implant were analyzed for the length of time to complete the expansion process (days)
Measure: Median (Full Range); unit: days
Units Other Than Participants: breasts
Arm/Group | AeroForm Tissue Expansion | Saline Tissue Expansion
Number analyzed (Participants) | 98 | 52
Number analyzed (breasts) | 142 | 82
days | 21 [6 to 169] | 46 [5 to 280]
Statistical Analysis 1: Comparison: AeroForm Tissue Expansion vs Saline Tissue Expansion; Test type: Superiority; p < 0.0001, Kaplan-Meier Log Rank test; Subjects not completing tissue expansion are censored in the analysis

ADVERSE EVENTS:
Time Frame: 1 year
Description: All AEs collected for the safety cohort (all subjects enrolled and procedure started). In the investigational arm (n=98 treated), the safety cohort includes one untreated subject in which the procedure was started but the device was not implanted due to intra-operative findings (positive nodes). Safety cohort for the investigation arm (n=99).
  AEs assessed by investigators for severity, seriousness and relationship to device or procedure.
  AEs coded to MedDRA standardized terms.
Arm/Group | AeroForm Tissue Expansion | Saline Tissue Expansion
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/52
Serious Adverse Events (participants affected / at risk) | 21/99 | 7/52
Other Adverse Events (participants affected / at risk) | 46/99 | 22/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AeroForm Tissue Expansion (N=99) | Saline Tissue Expansion (N=52)
Hematoma, Breast (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Post operative hematoma with return to the OR
Stroke, Mild (Nervous system disorders) | 1 (1) | 0 (0) — Mild Stroke, Admitted Overnight
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Fever with low wbc associated with chemotherapy
Red Breast Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Inflammation of the breast tissue
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Seroma with needle guided aspiration
Extrusion (General disorders) | 1 (1) | 1 (1) — Device extrusion through skin
Hematoma, Chest VAP Site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Hematoma after removal of Venous Access Port
Cellulitis (Infections and infestations) | 5 (6) | 2 (2) — Superficial Cellulitis of Breast
Wound Infection (Infections and infestations) | 1 (1) | 2 (2) — Wound Infection at the Surgical Site
Delayed Wound Healing (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) — Delayed wound healing, tissue necrosis
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Dehiscence (Separation) of the Incision
Erosion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Erosion of the skin overlying the expander
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Post operative pneumothorax
Deflation (General disorders) | 1 (1) | 1 (1) — Deflation
Under-Expansion (General disorders) | 1 (1) | 0 (0) — Under-Expansion
Over-Expansion (Product Issues) | 4 (5) | 0 (0) — Over-Expansion
Exposure (General disorders) | 1 (1) | 0 (0) — Exposed Tissue Expander
Muscle Disruption (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Disruption of Alloderm-Muscle Interface
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AeroForm Tissue Expansion (N=99) | Saline Tissue Expansion (N=52)
Pain (General disorders) | 10 (10) | 10 (10) — Subject Reported Pain
Delayed Wound Healing (Injury, poisoning and procedural complications) | 14 (14) | 3 (3) — Delayed Wound Healing / Tissue Necrosis,
Seroma (Injury, poisoning and procedural complications) | 14 (14) | 5 (5) — Seroma, Breast
Infection (Infections and infestations) | 8 (8) | 4 (4) — Post Op Wound Infection / Cellulitis

LIMITATIONS AND CAVEATS:
Device improvements occurred during the study with later subjects completing the study with a revised version of the device.

Results include all subjects treated in the study, regardless of device version.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No